CLINICAL TRIAL: NCT00699842
Title: A Phase I/II Optimal Dose Study of Lenalidomide in the Non-5q- LOW and INT-1 Risk MDS Patients
Brief Title: A Dose Range Finding Study of Lenalidomide in Non-5q Chromosome Deletion in Low and Intermediate Risk Myelodysplastic Syndrome (MDS) Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Administratively terminated per FDA recommendation
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07C.446; RV-MDS-PI-244 (Other: Celgene); 2007-31 (Other: CCRRC); JT 1238 (Other: JeffTrial Number)
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Myelodysplastic Syndrome; MDS; Low to Intermediate-1 MDS; Non-deletion 5q
Keywords: Myelodysplastic Syndrome; MDS; Low to Intermediate-1 MDS; Non-deletion 5q; Lenalidomide
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide will be given orally on day 1-21, followed by a 7day rest (28 day cycle). Cycles will be repeated every 28 days.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Dose Level Lenalidomide Schedule
  1. 15mg/day for d1-21 out of 28 days
  2. 20mg/day for d1-21 out of 28 days
  3. 25mg/day for d1-21 out of 28 days
  Other Names: Revlimid

SUMMARY:
Revlimid® (Lenalidomide) is indicated for a type of blood cancer, myelodysplastic syndrome (MDS), at 10mg for a specific type of myelodysplastic syndrome with a genetic abnormality called "deletion 5q" in Low and Intermediate-1 (INT-1) patients (staging system according to International Prognostic Scoring System (IPSS)). The purpose of this Phase I/II study is to determine the optimal dose of Revlimid® (Lenalidomide) in MDS Low and MDS INT-1 patients without deletion 5q by slowly increasing the dose while monitoring blood counts for safety evaluation as well as observe other adverse events. Efficacy will also be observed for the phase II portion of the study.

DETAILED DESCRIPTION:
There are little options for non deletion 5q Low and INT-1 patients. This study aims to find an early clinical signal for higher activity and better response with lenalidomide in patients with non deletion 5q Low and INT-1 MDS patients. Lenalidomide is an immunomodulatory agent. Thalidomide, the parent compound, has both immunomodulatory and anti-angiogenic properties which could confer anti-tumor and anti-metastatic efforts. Lenalidomide has been demonstrated to possess anti-angiogenic activity through inhibition of basic fibroblast growth factor (bFGF), vascular endothelial growth factor (VEGF) and tumor necrosis factor-alpha (TNF-alpha) induced endothelial cell migration (movement of cells in preparation to form new abnormal blood vessels for cancer cells), due at least in part to inhibition of Akt phosphorylation response to bFGF.

In addition, lenalidomide has a variety of immunomodulatory effects. Lenalidomide stimulates T cell proliferation, and the production of interleukin-2 (IL-2), IL-10 and interferon-gamma (IFN-gamma), inhibits IL-1 beta and IL-6 and modulated IL-12 production.

Although the exact anti-tumor mechanism of action of lenalidomide is unknown, a number of mechanisms are postulated for the activity of Lenalidomide in MDS.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. MDS patients who fulfill diagnostic criteria and classification by the IPSS Low or Int-1 categories according to cytogenetics, blood cytopenias and bone marrow blasts. See Appendix II.
5. All previous therapy such as azacitidine, decitabine, growth factors such as EPO (Procrit or Aranesp) and (Neupogen or Neulasta, Leukine, Neumega) or experimental therapy, must have been discontinued at least 4 weeks prior to treatment in this study.
6. ECOG performance status of 2 at study entry (see Appendix I).
7. Laboratory test results within these ranges:

   * Absolute neutrophil count 500/mm3
   * Platelet count 50,000 /mm3
   * Serum creatinine 2.0 mg/dL
   * Total bilirubin 1.5 mg/dL
   * AST (SGOT) and ALT (SGPT) 2 x ULN or 5 x ULN if hepatic metastases are present.
8. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix V: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods, AND also Appendix VI: Education and Counseling Guidance Document.
9. Disease free of prior malignancies for 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast

   * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. Concurrent use of other anti-cancer agents or treatments.
9. Known positive for HIV or infectious hepatitis, type A, B or C.
10. Myocardial infarction within 6 months prior to enrollment, or New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
11. History of thromboembolic disease within the past 6 months, regardless of anticoagulation

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Besa, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Associates in Hematology-Oncology, PC, Chester, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide (15mg); Lenalidomide (20mg); Lenalidomide (25mg): Lenalidomide will be given orally on day 1-21, followed by a 7day rest (28 day cycle). Cycles will be repeated every 28 days.
  Lenalidomide: Dose Level Lenalidomide Schedule
  1. 15mg/day for d1-21 out of 28 days
  2. 20mg/day for d1-21 out of 28 days
  3. 25mg/day for d1-21 out of 28 days
Period: Overall Study
Arm/Group | Lenalidomide (15mg) | Lenalidomide (20mg) | Lenalidomide (25mg)
Started | 3 | 5 | 0
Completed | 3 | 4 | 0
Not Completed | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide (15mg) | Lenalidomide (20mg) | Lenalidomide (25mg) | Total
Number analyzed (Participants) | 3 | 5 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.38 (20.06) | 65.98 (11.02) |  | 62.76 (14.29)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 2 | 3 |  | 5
  >=65 years | 1 | 2 |  | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 |  | 2
  Male | 3 | 3 |  | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 3 | 4 |  | 7
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0
  Not Hispanic or Latino | 1 | 2 |  | 3
  Unknown or Not Reported | 2 | 3 |  | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Determine CR, PR, and Rate of Stable Disease in MDS Patients
Description: Determine CR, PR, and rate of stable disease in MDS patients, IPSS Score LOW or INT-1 who do not have the 5q- cytogenetic abnormality according to the IWG criteria for response in >10mg doses of lenalidomide
Time Frame: 2 years
Arm/Group | Lenalidomide (15mg) | Lenalidomide (20mg) | Lenalidomide (25mg)
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Safety With Dose Escalation
Description: Safety (type, frequency, severity, and relationship of adverse events to study treatment) with dose escalation.
Time Frame: 2 years
Arm/Group | Lenalidomide (15mg) | Lenalidomide (20mg) | Lenalidomide (25mg)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Lenalidomide (15mg) | Lenalidomide (20mg) | Lenalidomide (25mg)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (15mg) (N=3) | Lenalidomide (20mg) (N=5) | Lenalidomide (25mg) (N=0)
Fatigue (General disorders) | 3 (4) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Numbness/tingling (Nervous system disorders) | 3 (4) | 3 (3) | 0 (0)
Hoarseness (General disorders) | 2 (2) | 0 (0) | 0 (0)
Swelling in legs (General disorders) | 1 (2) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (3) | 0 (0)
Awakening to urinate (Renal and urinary disorders) | 3 (4) | 3 (3) | 0 (0)
Pale skin (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Weakness (General disorders) | 2 (2) | 1 (1) | 0 (0)
Insomnia (General disorders) | 2 (2) | 2 (2) | 0 (0)
Post nasal drip (General disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle ache/pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Sore throat (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cough with sputum production (General disorders) | 2 (2) | 1 (1) | 0 (0)
Joint pain/stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0)
Problems with balance/dizziness (General disorders) | 1 (2) | 1 (2) | 0 (0)
Painful breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Elevated blood pressure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Swollen glands/lumps (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lack of energy/lack of motivation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Itching (General disorders) | 2 (2) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0)
Achiness under armpit (General disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in arm at injection site (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (General disorders) | 1 (2) | 1 (1) | 0 (0)
Sweats (General disorders) | 1 (1) | 2 (2) | 0 (0)
Sinus pain/congestion (General disorders) | 1 (1) | 2 (2) | 0 (0)
Dry eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (General disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (General disorders) | 1 (1) | 1 (1) | 0 (0)
Change in appetite (General disorders) | 0 (0) | 2 (2) | 0 (0)
Weight loss (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth/sores (General disorders) | 0 (0) | 1 (1) | 0 (0)
Shakiness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Memory changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Change in vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Itching of eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hip pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tired (General disorders) | 0 (0) | 1 (1) | 0 (0)
Red spots on leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Upset stomach (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Burning after urination (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dark urine (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swollen foot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Raised bumps on neck (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Lightheadedness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 0 (0) | 2 (2) | 0 (0)
Light flashes in right eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Pimple/boil (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Scattered rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in right hemithorax (General disorders) | 0 (0) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Shoulder pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Infection (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swollen abdomen (General disorders) | 0 (0) | 1 (1) | 0 (0)
Achiness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (General disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated as the objectives of this study have already been addressed in a larger study, and therefore the study is unlikely to yield any new information. The study closed before any data for the outcome measures was able to be collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes